CLINICAL TRIAL: NCT05520528
Title: Impact of Group Participation on Adults With Aphasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 274500
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Aphasia, Acquired; Stroke; Rehabilitation; Language Disorder, Acquired
MeSH Terms: conditions — Aphasia; Stroke; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reading Group (Experimental): All participants in this group will receive language intervention within weekly group sessions and independent tasks with emphasis on improving reading and writing skills among persons with aphasia.
  Interventions: Behavioral: Language intervention with group sessions and independent tasks with emphasis on improving reading and writing skills among persons with aphasia

INTERVENTIONS:
Behavioral: Language intervention with group sessions and independent tasks with emphasis on improving reading and writing skills among persons with aphasia — The participants will read through a designated book incrementally across multiple weeks at home and complete reading, writing, and discussion related to weekly readings in a group setting.

SUMMARY:
The purpose of the study is to examine the impact of group participation on adults with aphasia. Participants will complete a standard pre-and post-assessment of language abilities (speech, comprehension, reading, and/or writing). Then participants will attend 90-minute weekly reading group sessions during an academic semester.

DETAILED DESCRIPTION:
The objective of this research is to determine if attendance in groups positively impacts language skills, activity/participation, and/or quality of life in persons with aphasia.

This study will employ a university-clinic based outpatient group to administer language intervention. The specific aims of this study are to determine if group participation improves (1) life participation as measured by self-report questionnaires, (2) intervention-specific language skills as measured by treatment-related measures (e.g., reading comprehension and written expression), and (3) performance on non-treated language test scores as measured by a language assessment battery.

Participants will complete 4-5 individual testing sessions (e.g., initial assessment and pre-/post-testing), 7-12 group sessions (90-minute weekly reading group session), and 7-12 independent sessions at home (e.g., completion of weekly reading assignments).

The participants will read through a designated book incrementally across multiple weeks. The activities completed during the group sessions will focus on improving reading comprehension and written expression skills. Participants will read assigned passages at home and during the group sessions. Participants will complete a Copy and Recall Treatment (CART) worksheet independently to facilitate improvements in writing keywords related to the reading materials. CART involves copying target words and progresses to writing words from recall (Beeson, et al.). Participants will complete a reading comprehension worksheet and engage in discussion regarding the assigned book chapter.

Reading comprehension and written expression data will be collected and analyzed to compare the pre-treatment baseline performance from the first treatment session to the post-treatment performance from the last treatment session. Pre-and post-testing scores will be analyzed to investigate the change in scores across the 2-time points to determine the relative effectiveness of book club participation for improving reading comprehension, written expression, and life participation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pre-morbid proficient speaker of English
* Diagnosis of adult-onset aphasia
* Vision and hearing sufficient to complete assessments

Exclusion Criteria:

* No history of childhood speech or language difficulties
* No history of major psychiatric illness, cognitive impairment, or neurological disorders such as seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Reading Comprehension Battery for Aphasia-2 (RCBA-2; LaPointe & Horner, 1998) Scores | 1-week after intervention
  To determine if group participation improves intervention-specific language skills in reading comprehension by comparing baseline score to 1-week post-intervention score

SECONDARY OUTCOMES:
Communication Confidence Rating Scale for Aphasia (CCRSA; Babbitt & Cherney, 2010) | 1-week post-intervention
  To determine participant's feelings related to their communication. Participants rate their confidence on a scale from 0 to 100 for different communication-related activities. Baseline score will be compared to 1-week post-intervention score
Discourse Production Task | 1-week post-intervention
  Discourse analysis of participants producing monologic narratives (e.g., story retell, procedural explanation, picture sequence description, etc.). Baseline score will be compared to 1-week post-intervention score
Patient Reported Outcomes Measurement Information System (PROMIS) | 1-week post-intervention
  Selected PROMIS instruments (from cognitive, emotional, and social domains) will be used to measure satisfaction with and quality of life. Baseline score will be compared to 1-week post-intervention score.
Gray Oral Reading Test (GORT; Wiederholt & Bryant, 2012) | 1-week post-intervention
  To determine changes in oral reading and reading comprehension, baseline score will be compared to 1-week post-intervention score
Writing of Untrained Control Words (non-standardized). | 1-week post-intervention
  Writing untrained words that will be matched for frequency, length, and complexity with the CART trained words to measure generalization. Baseline score will be compared to 1-week post-intervention score

CONTACTS AND LOCATIONS:
Overall Officials: Dana Moser, Ph.D, Principal Investigator — University of Arkansas
Locations (1):
- UAM CHP Speech-Language and Hearing Clinic, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No